CLINICAL TRIAL: NCT06824428
Title: Can the Disease Subtype Affect the Pain Perception Threshold in Children Diagnosed With Attention Deficit Disorder With Hyperactivity?
Brief Title: The Pain Perception Threshold in Attention Deficit Disorder With Hyperactivity
Status: Completed | Type: Observational
Sponsor: Sultan 1. Murat State Hospital (Other Government)
Responsible Party: Principal Investigator, Alper Mengi, Associate Professor, Sultan 1. Murat State Hospital
Other Study IDs: 29/12/2024-Number:04
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pain Threshold; Attention Deficit Disorder With Hyperactivity (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Predominantly Inattentive: Patients diagnosed with inattentive subtype of attention deficit disorder with hyperactivity according to DSM-5 diagnostic criteria.
  Interventions: Other: Pain perception threshold
- Predominantly Hyperactive-Impulsive: Patients diagnosed with hyperactive-impulsive subtype of attention deficit disorder with hyperactivity according to DSM-5 diagnostic criteria.
  Interventions: Other: Pain perception threshold
- Inattentive and Hyperactive-Impulsive Combination: Patients diagnosed with mix subtype of attention deficit disorder with hyperactivity according to DSM-5 diagnostic criteria.
  Interventions: Other: Pain perception threshold

INTERVENTIONS:
Other: Pain perception threshold — The patients' pressure pain threshold will be evaluated with a manual pressure algometer (Baseline Dolorimtre®).The patients' pain perception thresholds will be measured bilaterally in the midfrontal region, the midpoint of the trapezius muscle, the lateral epicondyle, the midpoint of the web between the 1st and 2nd fingers, the greater trochanter, and the medial crease of the knee.

SUMMARY:
The aim of this study was to evaluate whether the disease subtype affects the presence of chronic pain and pain perception threshold in pediatric patients followed up with the diagnosis of attention deficit and hyperactivity disorder, and to evaluate the factors that may be related to pain perception threshold in disease subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with attention deficit and hyperactivity disorder according to DSM-5 diagnostic criteria
* Being between the ages of 6-17
* Being at a clinically normal mental level

Exclusion Criteria:

* Having verbal and visual communication problems
* Having a history of perinatal complications or physical head trauma
* Having comorbid psychiatric disorders other than oppositional defiant disorder and conduct disorder
* Known history of chronic physical and neurological disease (such as cerebral palsy, diabetes, epilepsy, autoimmune diseases, liver and kidney failure)
* Presence of substance or alcohol use disorder
* Having a genetic disorder diagnosis

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be selected from among those who apply to Edirne Sultan 1. Murat State Hospital Child and Adolescent Mental Health and Diseases polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-02-16 (Actual); Primary Completion 2025-12-26 (Actual); Study Completion 2025-12-26 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold | Baseline
  The pressure pain threshold will be assessed with a manual pressure algometer (Baseline Dolorimtre®). The patients' pain perception thresholds will be measured bilaterally in the midfrontal region, the midpoint of the trapezius muscle, the lateral epicondyle, the midpoint of the web between the 1st and 2nd fingers, the greater trochanter, and the medial crease of the knee. During the measurement, the 1.52 cm2 flat circular probe of the algometer will be placed on the relevant area and the pressure will be increased by 1 kg/second. Patients will be asked to express their pain by saying 'stop' or raising their hands when they feel slight discomfort. The value for each reference area will be obtained by calculating the arithmetic mean of the paired measurements.

SECONDARY OUTCOMES:
Presence of chronic pain | Baseline
  It will be questioned whether there has been continuous pain in any part of the body for at least 3 months.
Pain score | Baseline
  The patients' pain score will be evaluated with the Numerical Rating Scale (NRS). A 10 cm long horizontal straight line will be used in the NRS evaluation. Before the evaluation, the patient will be informed that a value of 0 represents no pain and a value of 10 represents the most severe pain felt to date. Patients will be asked to answer by considering the average of their pain over the last 3 days.
Duration of chronic pain | Baseline
  The duration of pain that has continued for at least 3 months in any part of the body will be questioned.
Sociodemographic data of patient | Baseline
  gender, age, height, weight, age of onset of complaints, duration of medication use, number of siblings, primary caregiver
Sociodemographic data of patient's parents | Baseline
  Age, occupation, education level and psychiatric disease history of mother and father

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Tiryaki, MD, Principal Investigator — Sultan 1. Murat State Hospital
Locations (1):
- Sultan 1. Murat State Hospital, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If requested, the data of the study will be shared by the researchers.